CLINICAL TRIAL: NCT06113692
Title: Clinical Course, Outcomes and Risk Factors of Myocarditis and Pericarditis Following Administration of mRNA- 1273 (ELASOMERAN)
Brief Title: A Study on the Clinical Course, Outcomes and Risk Factors of Myocarditis and Pericarditis After Moderna COVID-19 Vaccine
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Julius Clinical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P910
Record Dates: First submitted 2023-10-31; First posted 2023-11-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Myocarditis, Pericarditis
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna; Myocarditis; Pericarditis
MeSH Terms: conditions — Myocarditis; Pericarditis; Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; Spikevax bivalent zero omicron

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Moderna vaccination targeting SARS-CoV-2-exposed Case Cohort: All participants with myocarditis are selected among the participants who received at least 1 dose of Moderna vaccination targeting SARS-CoV-2. Cases are those participants who develop myocarditis or pericarditis any time during the follow-up after Moderna vaccination targeting SARS-CoV-2 vaccination.
  Interventions: Biological: mRNA-1273
- Myocarditis/Pericarditis Cohort: All participants with myocarditis and/or pericarditis with or without prior Moderna vaccination targeting SARS-CoV-2 exposure will be selected from the available databases.
  Interventions: Biological: mRNA-1273

INTERVENTIONS:
Biological: mRNA-1273 — intramuscular injection
  Other Names: Elasomeran; Imelasomeran; Davesomeran; Spikevax; Spikevax bivalent

SUMMARY:
The main goal of this study is to describe the clinical course, outcomes and risk factors for myocarditis and pericarditis associated with Moderna vaccination targeting SARS-CoV-2.

DETAILED DESCRIPTION:
This study will use an "Moderna vaccination targeting SARS-CoV-2 - exposed case cohort design" to assess the risk factors other than Moderna vaccination targeting SARS-CoV-2 vaccination for the development of myocarditis and pericarditis in Moderna vaccination targeting SARS-CoV-2 recipients, to understand which characteristics increase or decrease the risk for the development of myocarditis and pericarditis after Moderna vaccination targeting SARS-CoV-2 vaccination.

The second design "a myocarditis/pericarditis cohort study design" will be used to describe the prognostic factors for a severe clinical course in participants with myocarditis or pericarditis regardless of vaccination status. As most myocarditis and pericarditis cases are mild in disease severity, it is clinically relevant to identify the participants who are at increased risk for severe clinical outcomes (such as acute coronary syndrome, acute myocardial infarction, heart failure, atrial fibrillation/flutter, ventricular arrhythmias/cardiac arrest, pulmonary embolism or deep venous thrombosis, stroke outcomes, peripheral arterial embolism, hospital readmission, intensive care unit [ICU] admission or death) as early as possible in order to provide appropriate care in a timely manner. Therefore, information available at the onset of myocarditis or pericarditis could be used to predict the clinical course including long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* For the Elasomeran-Moderna vaccination targeting SARS-CoV-2-exposed case-cohort study, a cohort will be defined including participants of all ages with (1) at least one dose of Moderna vaccination targeting SARS-CoV-2 administered during the study period, (2) at least one year of enrolment in the applicable database prior to the index vaccine dose to allow for ascertainment of baseline covariables and potential risk factors, and (3) no myocarditis or pericarditis events within 6 months prior to Moderna vaccination targeting SARS-CoV-2 receipt. Myocarditis and pericarditis cases are defined when adjudication criteria similar to Centers for Disease Control and Prevention (CDC) case definition for probable or definite myocarditis or pericarditis is fulfilled.
* For the cohort study, participants will be included if they: (1) meet the adjudication criteria similar to the CDC case definition for probable or definite myocarditis or pericarditis, (2) have at least one year of enrolment in the applicable database prior to the index myocarditis or pericarditis event to allow for ascertainment of baseline covariates and potential risk factors, and (3) have not received a COVID-19 vaccine other than Moderna vaccination targeting SARS-CoV-2 within 30 days prior to the index myocarditis or pericarditis event.

Exclusion Criteria:

* Participants who have evidence of myocarditis or pericarditis in structured data (for example: ICD-10 codes) where review of clinical data is incompatible with adjudication criteria similar to CDC case definition for myocarditis or pericarditis will be described but will not be included as cases in primary analyses.
* In the Moderna vaccination targeting SARS-CoV-2-exposed case-cohort design, these non-confirmed myocarditis/pericarditis cases will be censored at the onset of the false positive myocarditis/ pericarditis diagnosis.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Information regarding participants is collected from multiple databases, utilizing routinely collected health and administrative data of four European countries: Denmark, Norway, Spain, and the United Kingdom. The study databases are representative of the source population in each country.
Sampling Method: Non-Probability Sample
Enrollment: 1169 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Myocarditis and/or Pericarditis within 30 Days After Moderna vaccination targeting SARS-CoV-2 | Up to 30 days post vaccination
Number of Participants With Severe Clinical Outcomes Within 30 Days After Onset of Myocarditis or Pericarditis | Up to 30 days after onset of myocarditis or pericarditis
  Clinical outcomes comprises of acute coronary syndrome, acute myocardial infarction, heart failure, atrial fibrillation/flutter, ventricular arrhythmias/cardiac arrest, pulmonary embolism or deep venous thrombosis, stroke outcomes, peripheral arterial embolism, hospital readmission, intensive care unit (ICU) admission or death.
Number of Participants With Long Term Clinical Outcomes After Onset of Myocarditis and/or Pericarditis | Up to 12 months

SECONDARY OUTCOMES:
Number of Participants With Severe Myocarditis or Pericarditis within 30 days After Moderna vaccination targeting SARS-CoV-2 | Up to 30 days post vaccination

CONTACTS AND LOCATIONS:
Locations (5):
- Aarhus University Hospital, Aarhus, Denmark
- University of Oslo, Oslo, Norway
- Spain (2):
  - IDIAP Jordi Gol, Barcelona
  - FISABIO, Valencia
- Drug Safety Research Unit (DSRU), Southampton, United Kingdom